CLINICAL TRIAL: NCT07326709
Title: A Randomized, Placebo-controlled, Double-blind Phase 3 Study to Evaluate the Efficacy, Safety and Tolerability of Votoplam in Participants With Huntington's Disease
Brief Title: A Study to Investigate the Efficacy, Safety and Tolerability of Votoplam in Participants With Huntington's Disease
Acronym: INVEST-HD
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHTT227A12301
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Huntington Disease
Keywords: HD; INVEST-HD; HTT227; VOTOPLAM; HUNTINGTON DISEASE; UHDRS; mHTT; NfL
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Votoplam (Experimental): Votoplam (blinded) taken orally, randomized in a 3:2 ratio (Votoplam: Placebo)
  Interventions: Drug: Votoplam (blinded)
- Placebo (Placebo Comparator): Placebo (blinded) taken orally, randomized in a 3:2 ratio (Votoplam: Placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Votoplam (blinded) — Votoplam (blinded) active treatment
  Other Names: HTT227
  Arms: Votoplam
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose is to assess safety and tolerability of votoplam and to determine whether votoplam slows disease progression in patients with early symptomatic Huntington's disease (HD) compared to the control arm.

HTT227 - current compound code (former code is PTC518 from PTC Therapeutics), HTT227 is Novartis code under Novartis sponsorship.

DETAILED DESCRIPTION:
This study will have a variable double-blind treatment duration of up to 36 months. As part of the study design, not every participant will complete 36 months of treatment.

The study consists of 3 periods:

* Screening Period: A period of up to 42-days to assess participants eligibility
* Double-blind Treatment Period: This period will have variable individual treatment duration, up to 36 months. The double-blind treatment period concludes when ≥50% patients complete Month 36. The maximum treatment duration for an individual participant is 36 months.
* Safety Follow-up Period: A period consisting of one safety follow-up visit, conducted on site or by phone call, for all participants not continuing treatment in the separate open-label extension study or discontinuing early. The visit/phone call will take place 30 days after End of Study (EOS)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consents must be obtained prior to participation in the study
* Ambulatory male or female participants between 21 to 70 years of age, inclusive, on the day of Informed Consent signature
* Genetically confirmed HD diagnosis with a cytosine-adenine-guanine (CAG) repeat length of 40 or above. Participants must have prior genetic confirmation and known CAG repeat length obtained prior to screening.
* Meets all of the following criteria:

  * UHDRS IS score ≥90
  * UHDRS TFC score = 13
  * UHDRS TMS score = 7-25, inclusive
  * CAP100 ≥ 70 Calculation: CAP = Age at study entry × (CAG length - 30) / 6.49

Exclusion Criteria:

* History of gene therapy or cell transplantation or any other experimental brain surgery for the treatment of HD
* Serologic evidence for active viral hepatitis as indicated by:

  * positive anti-HBc IgM
  * positive anti-HBc IgG confirmed by positive HBsAg and/or HBV DNA
  * positive HCV ab test confirmed by positive HCV RNA
  * Immunodeficiency diseases, including a positive human immunodeficiency virus (HIV) test result
* History or current diagnosis of ECG or cardiac abnormalities indicating significant risk of safety for participants such as:

  * Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second- or third-degree AV block without a pacemaker
  * History of familial long QT syndrome or known family history of Torsade de Pointes
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant from menarche until becoming post-menopausal, unless they have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral salpingectomy at least six weeks before taking study treatment. In the case of oophorectomy alone, the reproductive status of the woman needs to have been confirmed by follow-up hormone level assessment.

  o WOCBP are excluded unless they are using highly effective methods of contraception (failure rate < 1% per year) while taking study treatment and for 8 months after stopping study treatment.
* Pregnant or nursing (breastfeeding) women

Other protocol defined inclusion/exclusion criteria may apply

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-04-02 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in cUHDRS score | Baseline, Month 36
  The Composite Unified Huntingtons Disease Ratings Scale (cUHDRS) is an improved composite measure to assess multi-domain clinical progression in HD. The cUHDRS is a combined weighted score of measures of motor function (TMS), cognition (SDMT and SWRT) and overall functional capacity (TFC):
  cUHDRS = [(TFC-10.4)/1.9 - (TMS-29.7)/14.9 + (SDMT-28.4)/11.3 + (SWRT - 66.1)/20.1] + 10.
  In conjunction with one another, these measures provide a comprehensive, sensitive and specific tool for monitoring disease progression, with lower scores indicating more severe disease. cUHDRS score range from -8 to 25.

SECONDARY OUTCOMES:
Change from Baseline in UHDRS-TFC | Baseline, Month 36
  The UHDRS-Total Functional Capacity (TFC) focuses on the Investigator's assessment of the participant's capacity to perform a range of activities including occupation, finances, self-care, domestic chores and activities of daily living. The responses are derived from interview with the participant and/or companion, if applicable. Scores range from 0 to 13, with higher scores representing better functioning.
Change from Baseline in UHDRS-IS | Baseline, Month 36
  The UHDRS-Independence Scale (IS) measures a patient's overall level of functional independence in activities of daily living. It provides a single score ranging from 10 (total dependence/bedbound) to 100 (no special care needed) in intervals of 10, with higher scores indicating better functioning. Scores can also be assigned in increments of 5 for intermediate levels of function.
The time to decline in TFC score by at least one or IS score by at least 10 | Baseline to end of treatment up to 36 months
  The UHDRS-Total Functional Capacity (TFC) focuses on the Investigator's assessment of the participant's capacity to perform a range of activities including occupation, finances, self-care, domestic chores and activities of daily living. The responses are derived from interview with the participant and/or companion, if applicable. Scores range from 0 to 13, with higher scores representing better functioning.
  The UHDRS-Independence Scale (IS) measures a patient's overall level of functional independence in activities of daily living. It provides a single score ranging from 10 (total dependence/bedbound) to 100 (no special care needed) in intervals of 10, with higher scores indicating better functioning. Scores can also be assigned in increments of 5 for intermediate levels of function.
Change from Baseline in UHDRS-TMS | Baseline, Month 36
  The UHDRS-Total Motor Score (TMS) is the cumulative sum of the individual motor ratings obtained during the administration of the motor assessment portion of the UHDRS. It includes items related to eye movements, speech, limb movements (including hand taps and pronation-supination), dystonia, chorea, and gait/balance. Scores range from 0 to 124, with higher scores indicating greater motor impairment.
Change from Baseline in SDMT | Baseline, Month 36
  The Symbol Digit Modality Test (SDMT) is used to assess attention, working memory, psychomotor speed and visual perceptual processing. Participants are presented with a translation key of specific numbers paired with unique abstract symbols. Below the translation key is an array of symbols paired with empty spaces, the participant's task is to match the number for each symbol as quickly as possible in a given time frame. Scores are based on number of correctly paired items and range from 0 to 110, with higher scores representing better performance.
Change from Baseline in SWRT | Baseline, Month 36
  The Stroop Word Reading Test (SWRT) is a measure of processing and psychomotor speed. Participants are presented with a list or words (color names) printed in black ink and asked to read aloud as many words as possible within a set timeframe. Scores are based on the number of words read correctly and range from 0 to 60, with higher scores representing better performance.
Percent change from Baseline in blood mHTT protein | Baseline to steady state and up to 36 months in blood mHTT protein
  The mutant huntington protein (mHTT) which is detectable both in blood and cerebrospinal fluid (CSF), represents a reliable biomarker for HD due to its direct involvement in disease pathology.
  Blood mHTT is a direct product of the pathogenic HTT gene mutation and represents a proximal marker of Huntington's disease (HD) biology.
Change from Baseline in serum NfL | Baseline, Month 36
  Serum Neurofilament light chain NfL is a component of the neuronal cytoskeleton, released into CSF and blood after neuro-axonal damage, serving as a marker of neurodegeneration and disease progression in HD.
Incidence and severity of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) and TEAEs leading to participant withdrawal | Baseline to up to 36 months
  Number of participants with AEs and SAEs, including notable findings on physical examination, changes in vital signs, laboratory parameters, ECG, etc.

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com